CLINICAL TRIAL: NCT04696250
Title: Evaluation of Reporting of AdVerse Events Associated With AnTicAncer theRapy : an Observational and Retrospective Study Using the WHO Pharmacovigilance Database(AVATAR)
Brief Title: Evaluation of Reporting of AdVerse Events Associated With AnTicAncer theRapy (AVATAR)
Acronym: AVATAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: Pharmaco112020
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Antineoplastic Agents; Immunomodulating Agents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adverse Events associated with Antineoplastic and Immunomodulating Agents: Cases reported in the World Health Organization (WHO) and the French pharmacovigilance database of patients treated by anticancer drugs, with a chronology compatible with the drug toxicity
  Interventions: Drug: Antineoplastic and Immunomodulating Agents

INTERVENTIONS:
Drug: Antineoplastic and Immunomodulating Agents — Antineoplastic agents, endocrine therapy, immunostimulants and immunosuppressants drugs included in the ATC classification L

SUMMARY:
Anticancer drugs can lead to various adverse events. This study analyses reports of adverse events for treatment including Anatomical Therapeutic Chemical (ATC) classification L (antineoplastic agents, endocrine therapy, immunostimulants, and immunosuppressants drugs) in the World Health Organization's (WHO) global database of individual safety case reports (VigiBase).

DETAILED DESCRIPTION:
The investigators use VigiBase, the World Health Organization (WHO) database of individual safety case reports, to identify cases of adverse events following treatment with antineoplastic agents, endocrine therapy, immunostimulants or immunosuppressants drugs.

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the World Health Organization (WHO) database of individual safety case reports at the time of the extraction
* Adverse events reported were including in the MedDRA terms. The research could include the report with SOC, HGLT, HLT, or PT MedDRA terms
* Patients treated with Antineoplastic and immunomodulating agents included in the ATC L.

Exclusion Criteria:

* Chronology not compatible between the drug and the toxicity

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with Antineoplastic and immunomodulating agents
Sampling Method: Non-Probability Sample
Enrollment: 5000000 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events of antineoplastic and immunomodulating agents | Case reported in the World Health Organization (WHO) of individual safety case reports to January 1st 2025
  Identification and report of adverse event of antineoplastic and immunomodulating agents. The research could include the report with SOC, HGLT, HLT, or PT MedDRA terms

SECONDARY OUTCOMES:
Causality assessment of reported adverse events according to the WHO system | Case reported in the World Health Organization (WHO) of individual safety case reports to January 1st 2025
Description of the type of adverse event depending on the category of antineoplastic and immunomodulating agents | Case reported in the World Health Organization (WHO) of individual safety case reports to January 1st 2025
Description of the time from anticancer drug initiation and the occurrence of the adverse event | Case reported in the World Health Organization (WHO) of individual safety case reports to January 1st 2025
Description of the drug-drug interactions associated with adverse events | Case reported in the World Health Organization (WHO) of individual safety case reports to January 1st 2025
Description of the cancer for which the incriminated drugs have been prescribed | Case reported in the World Health Organization (WHO) of individual safety case reports to January 1st 2025
Description of the population of patients having adverse event | Case reported in the World Health Organization (WHO) of individual safety case reports to January 1st 2025

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandre Joachim, Caen, Basse Normandie, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] L'Orphelin JM, Da Silva A, Cabon J, Alexandre J, Dolladille C. Immune checkpoint inhibitor rechallenge after immune-related adverse events: a retrospective study from VigiBase update in 2024 looking for emergent safety signals. BMJ Open. 2024 Dec 3;14(12):e091708. doi: 10.1136/bmjopen-2024-091708. PMID 39627133